CLINICAL TRIAL: NCT00000612
Title: Soy Estrogen Alternative Study (SEA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 115; P01HL045666 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-11

CONDITIONS: Cardiovascular Diseases; Endometrial Hyperplasia; Heart Diseases; Menopausal Complaints; Uterine Diseases; Menopause
MeSH Terms: conditions — Cardiovascular Diseases; Endometrial Hyperplasia; Heart Diseases; Uterine Diseases | interventions — Estrogens, Conjugated (USP); Diet; Soybean Proteins; Dietary Supplements

INTERVENTIONS:
Drug: estrogens, conjugated
Behavioral: diet, soy proteins
Behavioral: dietary supplements

SUMMARY:
To conduct a three-armed trial assessing the effect of soy phytoestrogens on menopausal complaints, plasma lipids and lipoproteins, vaginal bleeding and endometrial proliferation, and health related quality of life.

DETAILED DESCRIPTION:
BACKGROUND:

The results of many studies indicate that estrogen replacement therapy (ERT) reduces the risk of coronary heart disease (CHD) in postmenopausal women. However, less than 9 percent of these women choose to take ERT because of unwanted side effects and concerns about increased risk of cancer associated with ERT. Therefore, alternative therapies are needed.

The isoflavonoids found in soy protein (specifically genistein) have many properties that may reduce the risk of coronary heart disease. These include favorable effects on plasma lipids and coronary artery vasomotion. Furthermore, genistein is a tyrosine kinase (TK) inhibitor with inhibitory effects on thrombin activity and TK receptor-linked mitogens that may be associated with atherogenesis and neointimal formation after angioplasty.

DESIGN NARRATIVE:

Randomized, double-blind, placebo-controlled. The women were randomized into one of three groups: placebo, conjugated equine estrogens, or soy supplementation. Primary endpoints were the impact on menopausal complaints such as hot flushes, mood lability, anxiety, sleep disturbances; effects on plasma lipids and lipoproteins, including lipoprotein (a); effects on vaginal bleeding and endometrial proliferation; changes in health-related quality of life. Secondary endpoints included: assessment of the impact of these interventions on the progression of carotid artery intimal medial wall thickening as assessed by B-mode ultrasonography; bone density and bone turnover; additional measures to monitor the compliance and safety of the intervention such as mammography, anticipated or known side effects of hormone replacement therapy, blood levels of genistein, and clinical outcomes such as hospitalizations, physician visits, and symptoms. The study ended in December, 1998.

The study was a subproject within a program project on coronary atherosclerosis in females, primarily monkeys. Dr. Thomas B. Clarkson was the P.I. The subproject dollars were estimated based on the CRISP dollars assigned to the study which were approximately 12 percent of the total program project dollars and were broken down as follows: FY 1996 - 219,254; FY 1997 - $217,000; FY 1998 - $221,000.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Perimenopausal/menopausal women, ages 45 to 55.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1996-01; Study Completion 1998-12 (Actual)

REFERENCES:
- [Background] Clarkson TB, Anthony MS, Williams JK, Honore EK, Cline JM. The potential of soybean phytoestrogens for postmenopausal hormone replacement therapy. Proc Soc Exp Biol Med. 1998 Mar;217(3):365-8. doi: 10.3181/00379727-217-44246. PMID 9492349